CLINICAL TRIAL: NCT05952804
Title: Immunoglobulin Replacement Therapy and Infectious Complications After CD19-Targeted CAR-T-Cell Therapy
Brief Title: IVIG for Infection Prevention After CAR-T-Cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Takeda (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG1123550; NCI-2023-04889 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20082 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA276040 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-07-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Solutions; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and study staff (except for site pharmacists) will be blinded to treatment arm assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (therapeutic immune globulin) (Experimental): Patients receive IGRT with IVIG within 14 days prior to CD19 CAR-T treatment. Patients then undergo CD19 CAR-T therapy. Patients receive IVIG monthly, starting 28 days after CD19 CAR-T therapy for 4 months in the absence of unacceptable toxicity. Patients also undergo blood sample collection throughout the study.
  Interventions: Biological: Immune Globulin Infusion (Human), 10% Solution; Biological: Anti-CD19 CAR T Cells Preparation; Procedure: Biospecimen Collection; Other: Survey Administration; Other: Electronic Health Record Review
- Arm II (normal saline) (Placebo Comparator): Patients receive placebo with normal saline IV within 14 days prior to CD19 CAR-T treatment. Patients then undergo CD19 CAR-T therapy. Patients receive normal saline monthly, starting 28 days after CD19 CAR-T therapy for 4 months in the absence of unacceptable toxicity. Patients also undergo blood sample collection throughout the study.
  Interventions: Biological: Anti-CD19 CAR T Cells Preparation; Other: Saline; Procedure: Biospecimen Collection; Other: Survey Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Biological: Immune Globulin Infusion (Human), 10% Solution — Given IV
  Other Names: GAMMAGARD LIQUID
  Arms: Arm I (therapeutic immune globulin)
Biological: Anti-CD19 CAR T Cells Preparation — Given CAR-T treatment
  Other Names: CD19-targeting CAR-T Cells
Other: Saline — Given IV
  Other Names: 7647-14-5; ISOTONIC SODIUM CHLORIDE SOLUTION; Sodium Chloride 0.9%
  Arms: Arm II (normal saline)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Survey Administration — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This phase II trial compares the effects of immunoglobulin replacement therapy with a placebo for preventing infectious complications in patients receiving CD19 chimeric antigen receptor (CAR)-T cell therapy. Hypogammaglobulinemia is a common complication in patients who receive CD19 CAR-T cell therapy. This is a condition in which the level of immunoglobulins (antibodies) in the blood is low and the risk of infection is high. Immunoglobulin replacement therapy works by replacing the body's immunoglobulin G (IgG) antibodies with donor blood product derived IgG antibodies that may help prevent infection. IgG antibodies are often depleted as a result of CAR-T therapy. Giving immunoglobulin replacement therapy may prevent infectious complications in patients receiving CD19 CAR-T cell therapy.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive immunoglobulin replacement therapy (IGRT) with intravenous immune globulin (IVIG) within 14 days prior to CD19 CAR-T-cell infusion. Patients then undergo CD19 CAR-T therapy. Patients receive IVIG monthly, starting 28 days after CD19 CAR-T therapy for up to 4 months in the absence of unacceptable toxicity, relapse of the underlying disease, or subsequent hematopoietic cell transplant. Patients also undergo blood sample collection throughout the study.

ARM II: Patients receive placebo with normal saline IV within 14 days prior to CD19 CAR-T treatment. Patients then undergo CD19 CAR-T-cell infusion. Patients receive normal saline monthly, starting 28 days after CD19 CAR-T therapy for up to 4 months in the absence of unacceptable toxicity, relapse of the underlying disease, or subsequent hematopoietic cell transplant. Patients also undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up monthly through up to 6 months after CD19 CAR-T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* For patients with medical incapacity or impaired consciousness such that they are not able to give fully informed voluntary consent, the subjects' legal representative must sign an institutional review board (IRB) approved informed consent document prior to the initiation of any screening or study-specific procedures
* Participants must be 18 years of age or older
* Participants will receive an Food and Drug Administration (FDA)-approved CD19-CAR T-cell product for the treatment of hematologic malignancies. Patients receiving an FDA-approved product are eligible even if the product is being administered as part of a clinical trial or expanded access program (e.g., product is 'out of specification'; concomitant anti-tumor treatment such as acalabrutinib)
* Serum total IgG < 600mg/dL within the prior three months
* SUBSEQUENT INFUSIONS: Received an FDA-approved CD19-CAR T-cell product for the treatment of hematologic malignancies

Exclusion Criteria:

* Primary congenital selective IgA deficiency
* Prior serious adverse event/s related to intravenous immune globulin (IVIG) administration
* Known serious allergy to any component of IVIG
* Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study or interfere with the patient's ability to participate for the full duration of the study or would put the patient at undue risk as judged by the investigator, such that it is not in the best interest of the patient to participate in this study
* SUBSEQUENT INFUSIONS: Ongoing symptoms of cytokine release syndrome (CRS) and/or immune effector cell-associated neurotoxicity syndrome (ICANS) meeting criteria for grade 3 or higher
* SUBSEQUENT INFUSIONS: Primary congenital selective IgA deficiency
* SUBSEQUENT INFUSIONS: Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study or interfere with the patient's ability to participate for the full duration of the study or would put the patient at undue risk as judged by the Investigator, such that it is not in the best interest of the patient to participate in this study
* SUBSEQUENT INFUSIONS: Receipt of additional therapy for persistence or relapse of the patient's primary malignancy
* SUBSEQUENT INFUSIONS: Receipt of bone marrow transplant (allogeneic or autologous)
* SUBSEQUENT INFUSIONS: Any serious adverse event (SAE), clinically significant adverse event (AE), severe laboratory abnormality, intercurrent illness, or other medical condition that indicates to the Investigator that continued participation is not in the best interest of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of serious bacterial infections in the modified intention-to-treat (mITT) population | From randomization through day 168 post chimeric antigen receptor (CAR) T-cell treatment (CARTx)
  Grade 2 or 3 bacterial infections. Only microbiologically confirmed infections will be included. Microbiological documentation of an infection consists of isolation of the pathogen by culture from a sterile (definite) or nonsterile (probable) site (if from a nonsterile site, the organism had to be clinically judged to be pathogenic). Will describe the number and type of infections in each study arm and calculate incidence rate estimates and 95% confidence intervals (CIs) for infections. Will compare serious bacterial infection incidence rates between study arms using negative binomial regression with an offset to account for days-at-risk. Will construct multivariable Cox proportional hazards models of time-to-first serious bacterial infection.

SECONDARY OUTCOMES:
Incidence rate of serious bacterial infections in ITT and per-protocol populations and of any serious infection or any infection after CD19 CARTx | From randomization through day 168 post CARTx
  Will use similar analytic approaches as in the primary outcome analysis to evaluate secondary outcomes (any serious infection, any infection) and all outcomes in pre-specified populations (mITT, per-protocol, ITT). Will explore outcomes restricted to early (days 0-28) and later (days 29-168) post-CARTx time periods. Plot cumulative incidence curves of time-to-first serious bacterial infection by study arm. Incidence rate ratios, hazard ratios (HR), and their 95% CIs will be reported. Will use one-sided testing to determine whether the rate of infections is significantly lower in the immunoglobulin replacement therapy (IGRT) versus placebo arms.
Levels of total IgG, IgG subclasses, and total Streptococcus (S.) pneumoniae IgG | From randomization through day 168 post CARTx
  Will graphically display mean total IgG levels, IgG subclasses, and S. pneumoniae IgG titers over time, stratified by study arm. Will use generalized estimating equations (GEE) models to compare means by randomization arm. Will test the association of each IgG metric as time-varying covariates with risk of subsequent infection (serious bacterial, any serious, any) at any time post-randomization and separately during early (days 0-28) and later (days 29-168) periods post-CARTx using Cox proportional hazard models. Model estimates will be presented as HRs with 95% CIs.
Health resource utilization (HRU) | Up to 6 months post CARTx
  Will describe HRU metrics by study arm (overall and by relationship to study drug infusion or infection). Will compute rates (per 1000 person-days) for each metric (e.g., days alive and out of the hospital, days of antibiotics, outpatient visits, emergency room visits, hospitalizations, adverse events) and compare between study arms using rate ratios with p-values and 95% CIs calculated by Poisson or negative binomial regression.
Incidence and severity of cytokine release syndrome (CRS) and/or immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 6 months post CARTx
  Will plot cumulative incidence curves, stratified by study arm, of any and grade >= 3 CRS, ICANS, or both, and compare hazard ratios using multivariable Cox proportional hazards models to adjust for stratification variables and potential confounders. To account for multiple comparisons, we will consider the Benjamini-Hochberg procedure for controlling the false discovery rate.
CAR T-cell expansion: Peak Plasma Concentration (Cmax) | Up to 6 months post CARTx
  Will display and compare between study arms the distribution of Cmax based on flow cytometry and quantitative polymerase chain reaction (qPCR) at weekly intervals between days 0 and 28 after CAR-T cell infusion using the Wilcoxon rank-sum test.
CAR T-cell expansion: area under the curve (AUC) | Up to 6 months post CARTx
  Will display and compare between study arms the area under the curve (AUC) 0-28 CAR-T cell values (log10 cells/uL) based on flow cytometry and quantitative polymerase chain reaction (qPCR) at weekly intervals between days 0 and 28 after CAR-T cell infusion using the Wilcoxon rank-sum test. The AUC 0-28 will be computed among log10-transformed CAR-T cell counts using a trapezoidal rule computational algorithm. Will use linear regression to test for differences in AUC 0-28 by study arm after adjusting for stratification variables (CAR-T cell product, site), disease burden (pre-lymphodepletion % bone marrow blasts; >= 5% versus < 5%), and other potential confounders.
CAR T-cell persistence | Up to 6 months post CARTx
  Will display the distribution of CAR-T cell values (log10 copies/ug deoxyribonucleic acid) per study arm based on monthly qPCR results and compare results using similar approaches as described for expansion. Timing of the loss of CAR-T cell persistence will be defined as the date of the first of two consecutive CAR-T cell values < 10 copies/ug. Will compute the cumulative incidence of loss of persistence and evaluate the association with study arm by day 168 using a Cox proportional hazards model including similar adjustment factors as previously described.
CAR T-cell phenotype and function | At day 14 post CARTx
  Compare CAR T-cell phenotype and function at day 14 after infusion between study arms. Cell subsets will be depicted using Uniform Manifold Approximation and Projection (UMAP), a dimension reduction technique to visualize and understand large, high dimensional datasets. Heatmaps will be created in R using the heatmap package to visualize differences in the proportion of patients with activated versus exhausted CAR-T cells and other select immune cell clusters, grouped for every marker and supervised by treatment arm. Will compare differences in absolute immune cell subset counts, the proportion of cell subsets with markers of activation versus exhaustion, and intracellular signaling (phospho-protein responses, stimulated and unstimulated) between study arms. Multivariable linear regression will be used to assess the relationship between treatment group and cell subset counts, as well as counts of activated versus exhausted cells, with adjustment for relevant confounders.
Immune cell subset phenotypes and functional makers | At 6 months post CARTx
  Compare all immune cell subset phenotypes and functional makers at the end of the study between study arms. Cell subsets will be depicted using UMAP, a dimension reduction technique to visualize and understand large, high dimensional datasets. Heatmaps will be created in R using the heatmap package to visualize differences in the proportion of patients with activated versus exhausted CAR-T cells and other select immune cell clusters, grouped for every marker and supervised by treatment arm. Will compare differences in absolute immune cell subset counts, the proportion of cell subsets with markers of activation versus exhaustion, and intracellular signaling (phospho-protein responses, stimulated and unstimulated) between study arms. Multivariable linear regression will be used to assess the relationship between treatment group and cell subset counts, as well as counts of activated versus exhausted cells, with adjustment for relevant confounders.
IgA and IgM levels | At 6 months post CARTx
  Compare IgA and IgM at end of study between study arms.
Health related quality of life (HRQOL) | From baseline up to 6 months post CARTx
  Compare HRQOL between study arms. Assessment of quality of life using the Patient Short Form-36 HRQOL electronic questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hill, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - City of Hope Cancer Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University (OHSU) Knight Cancer Institute, Portland, Oregon
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No